CLINICAL TRIAL: NCT05975138
Title: Marginal Bone Level Changes in Trans-gingival or Subcrestal Level Short Implants in the Atrophic Posterior Maxilla.
Brief Title: Trans-gingival or Subcrestal Short Implants Posterior Maxilla Bone Changes
Status: Completed | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Responsible Party: Sponsor
Other Study IDs: M2TRANS-SUB
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Alveolar Bone Resorption
Keywords: bone atrophy; dental implant; bone remodeling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- trans-gingival short implants: trans-gingival implant insertion in the posterior atrophic maxilla
  Interventions: Procedure: implant insertion
- subcrestal short implants: subcrestal implant insertion in the posterior atrophic maxilla
  Interventions: Procedure: implant insertion

INTERVENTIONS:
Procedure: implant insertion — a minimally invasive full-thickness flap will be raised in order to visualize the anatomy of the ridge. The vertical thickness of the supracrestal soft tissue will be measured and recorded. The preparation of the implant site will be performed with rotary burs and the bone quality will be recorded. An implant will be placed according to the manufacturer's recommendations. The length of the implant will be chosen in order to obtain a bicortical anchorage on the floor of the maxillary sinus
  Other Names: dental implant positioning

SUMMARY:
two groups of inserted implants: trans-gingival and under-bone level; difference in the marginal bone loss at six months from placement between the two groups of implant positioned in the posterior atrophic maxilla

DETAILED DESCRIPTION:
The inserted implants will be divided into two groups (group A: trans-gingival implants; group B: under bone level implants): a sample of 17 implants for each group was calculated to be necessary to detect a statistically significant difference in the marginal bone loss at six months from placement between the two groups (primary outcome) (alpha level set at 0.05 and statistical power at 80%) (Primer 6.0, Mc Graw-Hill, USA). The expected differences in marginal bone loss between groups (0.1 ±0.1 mm) were extrapolated from literature studies conducted on the topic10. Each center will treat 15 patients who need to insert implants in the posterior maxillary area, for a total of 45 implants, in order to compensate for any drop-outs.

Training and calibration session. Before the start of the study, a meeting will be held between all clinical centers to explain the surgical protocol, in order to ensure that clinical operators apply a standardized approach. A clinical operator for each center will receive written instructions regarding the evaluation of the experimental parameters in order to obtain repeatability in the collection of clinical parameters and in the compilation of the Case Report Form.

Screening stage.

All patients treated by the Clinical Centers are eligible to enter this study. Prior to enrollment, all patients will be required to sign an informed consent form to document that they understand the purpose of the study (including procedures, follow-up assessments, and potential risks involved). Patients will be allowed to ask questions related to this study and will be informed about alternative treatments.

Surgical procedure.

Presurgical planning will be performed with cone-beam computed tomography examination with or without the use of image reconstruction software.

After local anesthesia using articaine 4% with epinephrine 1:100,000, a minimally invasive full-thickness flap will be raised in order to visualize the anatomy of the ridge. The vertical thickness of the supracrestal soft tissue will be measured and recorded. The preparation of the implant site will be performed with rotary burs and the bone quality will be recorded. An implant (M2 Short, M2 Implants, Padova, Italy), 4 mm in diameter and 5, 6.5 or 7 mm in length, will be placed according to the manufacturer's recommendations (5 and 6.5 crestal placement; 7 subcrestal placement of 1 mm ). The length of the implant will be chosen in order to obtain a bicortical anchorage on the floor of the maxillary sinus.

Immediately after implant placement, an intraoral radiograph will be performed and an operator will record the implant stability values in the mesio-distal, disto-mesial, bucco-lingual and lingual-buccal directions. Dedicated disposable transducers and a measuring device will be used. The calibration of the instrument will be checked before and after each patient visit, using an implant fixed in a block of resin.

The flap will be sutured around the implant (one-stage protocol) with a non-absorbable monofilament, and an intraoral radiography with a centering device will be performed.

Patients will be prescribed antibiotics (amoxicillin/clavulanic acid 1 g 2 tablets/day from one day before surgery to five days after - clarithromycin 500 mg 1 tablet/day in allergic patients), NSAID (ibuprofen 600 mg as needed) and mouthwashes of chlorhexidine 0.2% lasting two minutes, three times a day.

The sutures will be removed 14 days after the surgery.

Postoperative recalls. After four months of healing, after periapical radiography and implant stability control , the final impression will be taken for the construction of the prosthetic product. The prosthetic rehabilitation will consist of single screw-retained ceramic crowns. Periapical radiographs will be performed upon delivery of the prosthetic product, after six months, one year, three and five years of prosthetic loading to evaluate the stability of the marginal bone.

Data analysis and retention. For each clinical center, a trained clinical operator and a clinical assistant will take care of data collection (filling in the case report form, performing periapical radiographs (on digital support) and measuring implant stability quotient values. Case report forms, radiographs and implant stability quotient measurements will be sent to the Coordination Centre, where trained operators will perform all measurements. The data will be transferred into a single electronic dataset for subsequent analysis. The examiners will not have been involved in the surgical and prosthetic phases and will proceed with the observation of the radiographs in a blind manner.

ELIGIBILITY:
Inclusion Criteria:

* 1) indications for an implant-prosthetic rehabilitation of a single edentulism in the upper posterior arch, on the basis of an accurate diagnosis and treatment planning;
* 2) the bone crest must be healed (at least six months after tooth loss);
* 3) residual bone crest width ≥6 mm;
* 4) presence of an available bone height between 4.5 and 8.5 mm on the floor of the maxillary sinus in the area of the planned implant insertion;
* 5) patient age >18 years;
* 6) the patient must not wear any type of removable prosthesis on the treated area;
* 7) the patient must be able to follow the study protocol;
* 8) written informed consent

Exclusion Criteria:

* 1) acute myocardial infarction in the last 2 months;
* 2) uncontrolled bleeding disorders;
* 3) uncontrolled diabetes (HBA1c > 7.5);
* 4) head/neck radiotherapy in the last 24 months;
* 5) immunocompromised patients, HIV positive or undergoing chemotherapy in the last 5 years;
* 6) current or past treatment with intravenous bisphosphonates;
* 7) psychological or psychiatric problems;
* 8) alcohol or drug abuse;
* 9) The local exclusion criterion is the presence of uncontrolled periodontal disease

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: people with an edentulous site in the posterior maxilla
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
marginal bone loss | six months
  millimeter of peri-implant bone resorption

SECONDARY OUTCOMES:
marginal bone loss | one year
  millimeter of peri-implant bone resorption

CONTACTS AND LOCATIONS:
Overall Officials: claudio stacchi, dr, Study Chair — International Piezoelectric surgery Academy
Locations (1):
- Piezosurgery Academy, Parma, Italy

IPD SHARING:
Plan to Share IPD: No
only after data elaboration

REFERENCES:
- [Background] Fan T, Li Y, Deng WW, Wu T, Zhang W. Short Implants (5 to 8 mm) Versus Longer Implants (>8 mm) with Sinus Lifting in Atrophic Posterior Maxilla: A Meta-Analysis of RCTs. Clin Implant Dent Relat Res. 2017 Feb;19(1):207-215. doi: 10.1111/cid.12432. Epub 2016 Jun 13. PMID 27295262
- [Background] Han HC, Lim HC, Hong JY, Ahn SJ, Han JY, Shin SI, Chung JH, Herr Y, Shin SY. Primary implant stability in a bone model simulating clinical situations for the posterior maxilla: an in vitro study. J Periodontal Implant Sci. 2016 Aug;46(4):254-65. doi: 10.5051/jpis.2016.46.4.254. Epub 2016 Aug 30. PMID 27588215
- [Background] Mezzomo LA, Miller R, Triches D, Alonso F, Shinkai RS. Meta-analysis of single crowns supported by short (<10 mm) implants in the posterior region. J Clin Periodontol. 2014 Feb;41(2):191-213. doi: 10.1111/jcpe.12180. Epub 2013 Nov 25. PMID 24266703